CLINICAL TRIAL: NCT00902824
Title: Phase I Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of TBC-M4 (MVA Based HIV Vaccine) Alone or in a Prime-Boost Regimen With ADVAX, DNA HIV Vaccine
Brief Title: Safety and Immunogenicity of TBC-M4, a MVA HIV Vaccine Alone or in a Prime-Boost Regimen With ADVAX DNA HIV Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI P002
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — delta inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Active Comparator): ADVAX at 0,1 and 2 months followed by TBC-M4 at 6 months
  Number of volunteers: 12
  Interventions: Biological: ADVAX
- Group B (Active Comparator): TBC-M4 at 0,1,6 months
  Number of volunteers: 12
  Interventions: Biological: TBC-M4
- Placebo (Placebo Comparator): Both Groups A and B will have 4 volunteers each (8 total) that will receive a placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ADVAX — Receive 4mg ADVAX at Months 0, 1, and 2 (Biojector), and receive boost of 5x10^7 pfu TBC-M4 (IM)
  Arms: Group A
Biological: TBC-M4 — Receive 5x10^7 pfu TBC-M4 (IM) at Months 0, 1, and 6.
  Arms: Group B
Other: Placebo — Group A (n=4) will receive the ADVAX placebo (formulation buffer) via Biojector.
  Group B (n=4) will receive the TBC-M4 placebo (formulation buffer) via IM.
  Arms: Placebo

SUMMARY:
This trial will study a prime-boost vaccine approach designed mainly to induce cell-mediated immune (CTL) responses.

DETAILED DESCRIPTION:
Two vaccine candidates will be used in two different prime-boost regimens: ADVAX (DNA) + TBC-M4 (MVA) and TBC-M4 (MVA) alone. Both these vaccines have already been tested in humans and both were found to be well tolerated and immunogenic. Approximately 32 volunteers (24 vaccine /8 placebo recipients) will be included in the study.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age on the day of screening and no greater than 50 years (i.e., had not reached his/her 51st birthday) on the day of first vaccination;
* Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study;
* In the opinion of the Principal Investigator or designee, has understood the information provided. Written informed consent needs to be given before any study-related procedures are performed;
* Willing to undergo HIV Testing, HIV counselling and receive HIV test results;
* If sexually active female, using an effective method of contraception (hormonal contraceptive; diaphragm; intrauterine device (IUD); condoms; anatomical sterility in self or partner) from screening until at least 4 months after last vaccination. All female volunteers must be willing to undergo urine pregnancy tests at time points as indicated in the Schedule of Procedures (Appendix A);
* If sexually active male, willing to use an effective method of contraception (such as condoms, anatomical sterility) from the day of enrolment until at least 4 months after the last vaccination;
* Willing to forgo donations of blood, sperm, eggs, bone marrow or organs during the study.

Exclusion Criteria:

* Confirmed HIV-1 or HIV-2 infection;
* High-risk behaviour for HIV infection which is defined as (Within 6 months before vaccination, the volunteer has):

  * Had unprotected vaginal or anal sex with a known HIV infected person or a casual partner (i.e., no continuing established relationship)
  * Engaged in sex work for money or drugs
  * Substance abuse/use injection drugs
  * Acquired a sexually transmitted disease (STD) (e.g., gonorrhoea, chlamydia, syphilis, Trichomonas vaginalis, and symptomatic herpes genitalis)
  * Having a high-risk partner either currently or within the previous 6 months
* Any clinically significant abnormality on history or examination including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids, immunosuppressive, antiviral, anticancer, or other medications considered significant by the investigator within the previous 6 months; (Note: use of inhaled steroids for asthma and use of topical steroids for localized skin conditions will not exclude a volunteer from participation.)
* Any clinically significant acute or chronic medical condition that is considered progressive or in the opinion of the investigator would make the volunteer unsuitable for the study;
* Any of the following abnormal laboratory parameters listed below:

  * Haemoglobin <10.0 g/dL
  * Absolute Neutrophil Count (ANL): <1,000/mm3
  * Absolute Lymphocyte Count (ALC): <600/mm3
  * Platelets: <100,000/mm3
  * Creatinine: >1.3 x ULN
  * AST: >2.5 x ULN
  * ALT: >2.5 x ULN
  * Cardiac Troponin I: > ULN
  * Urinalysis: Abnormal dipstick confirmed by microscopy:

    * blood = 3+ or more (not due to menses)
    * protein = 3+ or more
    * leucocytes = 3+ or more
* Confirmed diagnosis of hepatitis B (HBsAg), hepatitis C (HCV antibodies), or active syphilis;
* If female, pregnant or planning a pregnancy within 4 months after last vaccination; or lactating;
* Receipt of live attenuated vaccine within the previous 60 days (live attenuated flu vaccine within 14 days) or planned receipt within 60 days after vaccination with Investigational Product or receipt of other vaccine within the previous 14 days or planned receipt within 14 days after vaccination with Investigational Product;
* Receipt of blood transfusion or blood products within the previous 6 months.
* Participation in another clinical study of an investigational product currently, within the previous 3 months or expected participation during this study;
* Receipt of another investigational HIV vaccine in the last 6 years (note: receipt of an HIV vaccine placebo will not exclude a subject from participation if documentation is available to the study site and the IAVI Medical Monitor gives approval);
* History of severe local or systemic reactogenicity to vaccines or history of severe allergic reactions;
* Major psychiatric illness including any history of schizophrenia or severe psychosis, bipolar disorder requiring therapy, suicidal attempt or ideation in the previous 3 years;
* Smallpox vaccination within the previous 3 years;
* ECG with clinically significant findings or features that would interfere with the assessment of myopericarditis, including but not limited to:

  * Conduction disturbance (atrio-ventricular or intra-ventricular conduction, left or right bundle branch block, AV block of any degree, or QTc prolongation)
  * Repolarization (ST segment or T wave) abnormality
  * Significant atrial or ventricular arrhythmia
  * Frequent atrial or ventricular arrhythmia
  * Frequent atrial or ventricular ectopy (e.g., frequent premature atrial contractions, two premature ventricular contractions in a row)
  * ST elevation consistent with ischemia
  * Evidence of past or evolving myocardial infarction (heart attack).
* History of, or known active cardiac disease, including but not limited to:

  * Previous myocardial infarction
  * Angina pectoris
  * Congestive heart failure
  * Valvular heart disease, including mitral valve prolapse
  * Cardiomyopathy
  * Pericarditis
  * Stroke or transient ischemic attack
  * Chest pain or shortness of breath with activity (such as walking up stairs)
  * Other heart conditions under the care of a doctor.
* Have 3 or more of the following risk factors:

  * High blood pressure diagnosed by a doctor
  * High blood cholesterol diagnosed by a doctor
  * Diabetes
  * High blood sugar diagnosed by a doctor
  * First degree relative (e.g., mother, father, brother, sister) who had a heart condition before the age of 50
  * Smoke cigarettes now.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety of TBC-M4 alone or in a prime-boost regimen with ADVAX | 12 months
  Safety and tolerability of TBC-M4 alone (given im) or in a prime-boost regimen with ADVAX (administered by Biojector)

SECONDARY OUTCOMES:
Immunogenicity of TBM-M4 alone or in a prime-boost regimen with ADVAX | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian Gazzard, MD, Principal Investigator — St. Stephen's Centre
Locations (1):
- St Stephen's Centre Chelsea and Westminster Hospital, London, London, United Kingdom

REFERENCES:
- See also: International AIDS Vaccine Initiative — http://www.iavi.org